CLINICAL TRIAL: NCT00723827
Title: Temodal (Temozolomide) Post Marketing Surveillance Protocol
Brief Title: Temodal (Temozolomide) Post Marketing Surveillance Protocol (Study P05557AM2)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05557
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2013-01-08 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Glioblastoma; Glioma; Astrocytoma
MeSH Terms: conditions — Glioblastoma; Glioma; Astrocytoma | interventions — Temozolomide; Radiotherapy; Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Participants with newly diagnosed glioblastoma multiforme (treat with temozolomide & radiotherapy) or participants with malignant glioma, such as glioblastoma multiforme or anaplastic astrocytoma, showing recurrence or progression after standard therapy (treat with temozolomide).
  Interventions: Drug: Temozolomide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Temozolomide — Administration of temozolomide based on the product labeling.
  Other Names: Temodal; Temodar; SCH 052365; MK-7365
Radiation: Radiotherapy — Radiotherapy given concomitantly with temozolomide for newly diagnosed glioblastoma multiforme.
  Other Names: Radiation therapy; irradiation

SUMMARY:
The purpose of this surveillance is to evaluate the postmarketing safety and efficacy of Temodal capsule (temozolomide) under actual conditions of use, and to understand some of the following points that are in question and doubt:

* Incidence of adverse events under actual conditions of use (Serious and Nonserious Adverse Events);
* Adverse Drug Reactions not shown in the directions for use (will be stated as Unexpected Adverse Reaction);
* Adverse Event caused by misuse, abuse, or drug interactions;
* Other information concerned with safety or efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are prescribed with temozolomide by local labeling:

  * participants with newly diagnosed glioblastoma multiforme;
  * participants with malignant glioma, such as glioblastoma multiforme or anaplastic astrocytoma, showing recurrence or progression after standard therapy.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with newly diagnosed glioblastoma multiforme.
  Participants with malignant glioma, such as glioblastoma multiforme or anaplastic astrocytoma, showing recurrence or progression after standard therapy.
Sampling Method: Probability Sample
Enrollment: 682 (Actual)
Dates: Start 2008-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Participants with newly diagnosed glioblastoma multiforme (treat with temozolomide & radiotherapy) or participants with malignant glioma, such as glioblastoma multiforme or anaplastic astrocytoma, showing recurrence or progression after standard therapy (treat with temozolomide).
  Temozolomide : Administration of temozolomide based on the product labeling.
  Radiotherapy : Radiotherapy given concomitantly with temozolomide for newly diagnosed glioblastoma multiforme.
Period: Overall Study
Arm/Group | All Participants
Started | 682
Completed | 682
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 682
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.57 (13.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 297
  Male | 385
Region of Enrollment [Number; unit: participants]
  Korea, Republic Of | 682

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of vaccine, whether or not considered related to the medicinal product.
Time Frame: Complete study duration & 30 days after completion (up to approximately 7.5 months)
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 682
participants | 324

2. Primary Outcome: Number of Participants Experiencing Unexpected Adverse Drug Reactions (ADRs)
Description: An unexpected ADR was defined as an adverse reaction, whose nature, severity, specificity, or outcome is not consistent with the term or description used in the applicable product information.
Time Frame: Complete study duration & 30 days after completion (up to approximately 7.5 months)
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 682
participants | 49

3. Primary Outcome: Number of Temozolomide Misuse or Abuse Events
Description: Drug abuse was defined as the use of the study drug for a non-therapeutic effect.
  Misuse was defined as use of the study medication in a way that was not prescribed.
Time Frame: Complete study duration & 30 days after completion (up to approximately 7.5 months)
Measure: Number; unit: Events
Arm/Group | All Participants
Number analyzed (Participants) | 682
Events | 1

4. Primary Outcome: Number of Temozolomide Drug Interactions
Description: Drug interaction was defined as a chemical or physiological reaction that can occur when two different drugs are taken together.
Time Frame: Complete study duration & 30 days after completion (up to approximately 7.5 months)
Measure: Number; unit: events
Arm/Group | All Participants
Number analyzed (Participants) | 682
events | 5

5. Primary Outcome: Efficacy: Number of Participants Experiencing Complete Response (CR), Partial Response (PR), or Stable Disease(SD)
Description: The response ratings were based on the judgment of the investigator.
Time Frame: Complete study duration (up to approximately 6.5 months)
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 682
participants
  CR | 82
  PR | 143
  SD | 322

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 103/682
Other Adverse Events (participants affected / at risk) | 132/682
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=682)
EOSINOPHILIA (Blood and lymphatic system disorders) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (4)
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2)
CARDIAC ARREST (Cardiac disorders) | 2 (2)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1)
VISION BLURRED (Eye disorders) | 1 (1)
VISUAL IMPAIRMENT (Eye disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 3 (3)
ASTHENIA (General disorders) | 3 (3)
CHEST DISCOMFORT (General disorders) | 1 (1)
CHILLS (General disorders) | 1 (1)
CONDITION AGGRAVATED (General disorders) | 2 (2)
DISEASE PROGRESSION (General disorders) | 17 (17)
FACE OEDEMA (General disorders) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1)
PYREXIA (General disorders) | 7 (7)
HEPATITIS (Hepatobiliary disorders) | 1 (1)
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
CENTRAL NERVOUS SYSTEM INFECTION (Infections and infestations) | 1 (1)
HEPATITIS B (Infections and infestations) | 1 (1)
LOCALISED INFECTION (Infections and infestations) | 1 (1)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 11 (11)
SEPSIS (Infections and infestations) | 2 (2)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Renal and urinary disorders) | 2 (2)
WOUND INFECTION (Infections and infestations) | 3 (3)
RADIATION NECROSIS (Injury, poisoning and procedural complications) | 2 (2)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 (2)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (4)
OXYGEN SATURATION DECREASED (Investigations) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTASES TO SPINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NEOPLASM RECURRENCE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
BRAIN OEDEMA (Nervous system disorders) | 4 (4)
CEREBRAL CYST (Nervous system disorders) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1)
CONVULSION (Nervous system disorders) | 9 (11)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (2)
DYSARTHRIA (Nervous system disorders) | 2 (2)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 5 (5)
HYDROCEPHALUS (Nervous system disorders) | 5 (5)
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 1 (1)
MYELOPATHY (Nervous system disorders) | 1 (1)
PARTIAL SEIZURES (Nervous system disorders) | 2 (2)
SOMNOLENCE (Nervous system disorders) | 2 (2)
STUPOR (Nervous system disorders) | 2 (2)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2 (2)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2 (2)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 3 (3)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=682)
NAUSEA (Gastrointestinal disorders) | 82 (101)
VOMITING (Gastrointestinal disorders) | 54 (64)
DECREASED APPETITE (Metabolism and nutrition disorders) | 46 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution has the right to publish/present the study results. The institution agrees not to publish/present any interim results of the Study without the Sponsor's prior written consent. The institution further agrees to provide the Sponsor 30 days written notice prior to submission. The Sponsor has the right to review and comment. If the parties disagree, the institution agrees to meet with the Sponsor, prior to submission, to discuss and resolve any such issues or disagreement.